CLINICAL TRIAL: NCT01530334
Title: A Phase II Open Label, Multicentre, Single Arm Study to Characterise the Efficacy, Safety and Tolerability of Gefitinib 250 mg (IRESSA) as 3rd Line Treatment Re-challenge in Patients, Who Have Epidermal Growth Factor Receptor (EGFR) Mutation Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) and Who Responded to Gefitinib in 1st Line and Progressed After 2nd Line Chemotherapy
Brief Title: Iressa Re-Challenge in Advanced NSCLC EGFR M+ Patients Who Responded to Gefitinib USed as 1st Line or Previous Treatment
Acronym: ICARUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7913L00138; EUDRACT n 2011-005157-31
Record Dates: First submitted 2012-01-31; First posted 2012-02-09 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gefitinib

ARMS (1):
- open label single arm with Gefitinib 250MG once daily (Experimental): Gefitinib 250 mg/day open label until progression disease / toxicity / consent withdrawal
  Interventions: Drug: Gefitinib 250mg

INTERVENTIONS:
Drug: Gefitinib 250mg — Gefitinib 250mg once daily
  Other Names: Iressa

SUMMARY:
the primary objective is to characterise the impact of gefitinib on the Response Evaluation Criteria in Solid Tumours (RECIST) based assessments; objective response rate (ORR ; confirmed complete response(CR) or partial response (PR)) and disease control rate (DCR; confirmed complete response(CR) or partial response (PR) or stable disease (SD)) in patients with EGFR M+ NSCLC

DETAILED DESCRIPTION:
A phase II Open Label, Multicentre, Single Arm Study to Characterise the Efficacy, Safety and Tolerability of Gefitinib 250 mg (IRESSA�) as 3rd line treatment re-challenge in Patients, who have Epidermal Growth Factor Receptor (EGFR) Mutation Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) and who responded to gefitinib in 1st line and progressed after 2nd line chemotherapy

ELIGIBILITY:
Inclusion Criteria at screening (Visit 1) and at Start of Study Treatment (Visit 2):

* Provision of informed consent prior to any study specific procedures.
* Histologically or cytologically confirmed NSCLC with an activating sensitising EGFR TK mutation as it was determined before starting the first gefitinib treatment by using a well-validated and robust methodology: adenocarcinoma, including Bronchoalveolar Carcinoma (BAC), squamous cell carcinoma, large cell carcinoma, adenosquamous carcinoma or undifferentiated carcinoma or not-otherwise specified NSCLC.

  * Female or male patients aged 18 years or over with Locally advanced or metastatic stage IIIB/IV disease, not suitable for therapy of curative intent or stage IV (metastatic) disease, eligible for gefitinib re-challenge treatment for NSCLC who have already received gefitinib with a documented complete (CR) or partial response (PR) or stable disease (SD) >12 weeks as the best response to their 1st gefitinib treatment and progressing during or after a subsequent anti-cancer therapy (excluding EGFR-TKIs) treatment, including but not limited to doublet platinum based chemotherapy or docetaxel monotherapy or pemetrexed monotherapy.
  * Measurable disease defined as at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with spiral CT or MRI and which is suitable for accurate repeated measurements.
  * WHO / ECOG / Zubrod performance status 0-2.

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of the product
* Prior EGFR TKIs except gefitinib followed by subsequent anti-cancer treatment (including chemotherapy and excluding EGFR-TKIs).

Previous adjuvant chemotherapy is allowed. Prior surgery or radiotherapy must be completed more than 6 months before start of study treatment. Palliative radiotherapy must be completed at least 4 weeks before start of study treatment with no persistent radiation toxicity.

* Progression disease or stable disease (SD) <12 weeks as best response to the 1st line treatment with gefitinib
* Not progressing during or after the last anti-cancer treatment.
* Considered to require radiotherapy to the lung at the time of study entry or in the near future
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease
* Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline
* Insufficient lung function as determined by either clinical examination or an arterial oxygen tension (PaO2) of < 70 Torr
* Known or suspected brain metastases or spinal cord compression, unless treated with surgery and/or radiation and stable without steroid treatment for at least 4 weeks prior to the first dose of study medication
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Concomitant use of known CYP 3A4 inducers such as phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort
* Pregnancy or breast-feeding
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (eg, unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Life expectancy of less than 12 weeks

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Riggi, MD MEDICAL DIRECTOR, Study Director — AstraZeneca SpA, Medical Dept., Basiglio, ITALY; Filippo Marinis, MD, Principal Investigator — S.Camillo-Forlanini High Specialization Hospitals, Rome, ITALY; Silvia Ferrari, MD, Study Director — AstraZeneca SpA, Medical Dept., Basiglio, ITALY
Locations (24):
- Italy (24):
  - Research Site, Alessandria
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cona
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Lecce
  - Research Site, Macerata
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Pordenone
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Treviso
  - Research Site, Udine
  - Research Site, Verona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 61 patients were enrolled from July 2012 to July 2014 from 25 medical clinics across Italy: of these, 59 received gefitinib.
Pre-assignment Details: The study foresees a screening period of 28 days where the investigator had to obtain signed informed consent from the potential patient before any study specific procedures are performed, and determine patient eligibility. At the end of the screening period the patient started the treatment with gefitinib
Groups:
- Gefitinib: 250 mg/die, oral
Period: Overall Study
Arm/Group | Gefitinib
Started | 61
Completed | 10
Not Completed | 51
Not completed — Adverse Event | 3
Not completed — unknown reason | 1
Not completed — Progressive disease | 47

BASELINE CHARACTERISTICS:
Population: The overall number of patients was 61 (FAS population). FAS population was defined as all screened patients enrolled in the study
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 16
Race/Ethnicity, Customized [Number; unit: Participants] — All patients were Caucasian (61, 100%)
  Participants
    White | 61

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective Response Rate is the sum of Complete response (CR) and Partial Response (PR) response.
  Evaluated by recist criteria v 1.1., for target lesions and assesed by CT or MRI: Complete Response (CR), Disapperance of all target lesions; Partial Response (PR),>=30% decrease in the sum of longest diamteter of target lesions; Objective response rate (RR)=CR+PR
Time Frame: every 6 weeks after the Start of Study Treatment until objective disease progression or time of data cut off (6 months after the last patient has started study treatment)
Population: Analysis performed both in the FAS population (i.e. all enrolled patients into the study) and in EFS population (i.e. all screened patients who entered and received at least one dose of study agent)
Measure: Number; unit: Patients
Units Other Than Participants: partecipants
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
Number analyzed (partecipants) | 61
Patients | 3

2. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is the sum of patients with a best visit response of Complete Response, Partial Response or Stable Desease Objective Response Rate is the sum of Complete response (CR) and Partial Response (PR) response.
  Evaluated by recist criteria v 1.1., for target lesions and assesed by CT or MRI: Complete Response (CR), Disapperance of all target lesions; Partial Response (PR),>=30% decrease in the sum of longest diamteter of target lesions, Stable Desease (SD) defined as no progression for>= 6 weeks. Objective response rate (RR)=CR+PR
Time Frame: as for outcome 1
Population: CBR was analyzed both on FAS and EFS population
Measure: Number; unit: Patients
Units Other Than Participants: Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
Patients | 32 [40.2 to 64.5]

3. Secondary Outcome: Progression Free Survival
Description: Progression free Survival was calculated as the time from the first dose of gefitinib study treatment until the date of (i) progression or (ii) death from any cause in the absence of progression.
Time Frame: as for outcome 1
Population: PFS was analysed on FAS and EFS population
Measure: Median (95% Confidence Interval); unit: Days
Units Other Than Participants: Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
Days | 84 [74 to 94]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated as the time from the first dose until the day of death from any cause. Any patient not known to have died at the time of data analysis was censored at the time of the last follow-up date.
Time Frame: every 6 weeks after the Start of Study Treatment until death or time of data cut off (6 months after the last patient has started study treatment)
Population: Analysis conducted both in FAS and EFS population
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
days | 311 [268 to 431]

5. Secondary Outcome: Treatment Duration With Gefitinib
Description: Treatment duration was calculated from the date of the first to the date of the last intake.
Time Frame: every 6 weeks after the Start of Study Treatment until discontinuation of drug or time of data cut off (6 months after the last patient has started study treatment)
Population: Analysis performed on EFS & FAS population
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
days | 108 [92 to 169]

6. Secondary Outcome: Time to Worsening of Disease Related Symptoms
Description: Time to worsening of disease related symptoms (LCS) Time to worsening of disease-related symptoms based on FACT-L LCS was defined as the interval from the date of enrollment to the first visit response of 'worsened' without a subsequent response of 'improved' or 'no change' within 21 days (or to the last assessment), death due to any cause, or early discontinuation from the study. Time to worsening was censored at the last non-missing assessment visit if the worsening was not observed.
Time Frame: every 6 weeks after the Start of Study Treatment until the worsening of desease related symptoms or time of data cut off (6 months after the last patient has started study treatment)
Population: Analysis performed on EFS & FAS population
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 61
days | 93 [71 to 109]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse Events and Serious Adverse Events were collected from the time of screening informed consent throughout the treatment period, until 30 days after discontinuation of gefitinib treatment. Adverse events were based on sign and symptoms reported by the patients and on examinations and test
Arm/Group | Gefitinib
Serious Adverse Events (participants affected / at risk) | 10/58
Other Adverse Events (participants affected / at risk) | 42/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib (N=58)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib (N=58)
Diarrohea (Gastrointestinal disorders) | 16 (21)
Vomiting (Gastrointestinal disorders) | 9 (11)
Nausea (Gastrointestinal disorders) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 9 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Skin toxicity (Skin and subcutaneous tissue disorders) | 3 (5)
Asthenia (General disorders) | 5 (8)
Chest pain (General disorders) | 5 (5)
Fatigue (General disorders) | 5 (5)
Pyrexia (General disorders) | 5 (6)
General physical health deterioration (General disorders) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Folliculitis (Infections and infestations) | 3 (3)
Paronychia (Infections and infestations) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Conjunctivitis (Eye disorders) | 5 (12)
Hypertension (Vascular disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other